CLINICAL TRIAL: NCT00658320
Title: A 12-month, Multicenter, Randomized, Open-label Study to Investigate Efficacy and Safety of Concentration Controlled Everolimus With Reduced Dose Cyclosporine A Versus Mycophenolate Mofetil With Standard Dose Cyclosporine A in de Novo Renal Transplant Adult Recipients Treated With Basiliximab and Corticosteroids
Brief Title: Concentration Controlled Everolimus With Reduced Dose Cyclosporine Versus Mycophenolate Mofetil With Standard Dose Cyclosporine in de Novo Renal Transplant Adult Recipients Treated With Basiliximab and Corticosteroids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRAD001A1202; NCT00856466 (obsolete NCT alias)
Record Dates: First submitted 2008-04-10; First posted 2008-04-15 (Estimated); Results first posted 2011-09-14 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-05

CONDITIONS: Kidney Transplantation
Keywords: Renal transplantation; everolimus; mycophenolate mofetil; cyclosporine; corticosteroid; basiliximab; Banff diagnosis; Acute rejection; Therapeutic drug monitoring (TDM); de novo renal transplant recipient
MeSH Terms: interventions — Everolimus; Mycophenolic Acid; Basiliximab; Cyclosporine; Adrenal Cortex Hormones

ARMS (2):
- Everolimus + Reduced dose of cyclosporine (Experimental): An initial everolimus dose of 0.75 mg orally twice daily (1.5 mg/day) was administered 24-36 hours from reperfusion after transplantation and dose adjustments based on everolimus trough level (target trough level 3-8 ng/mL). Reduced dose of cyclosporine was initiated either pre-transplantation or within 24 hours after transplantation following the local regimen. Patients were treated with antibody induction therapy using 20 mg basiliximab two hours prior to transplant and 20 mg basiliximab 4 days post transplant or according to local practice. Corticosteroids were administered according to local practice. Patients were treated for 12 months in the core study and 12 months in the extension study. Everolimus was available after 24 months for compassionate use.
  Interventions: Drug: Everolimus; Drug: Basiliximab; Drug: Cyclosporine A; Drug: Corticosteroid
- Mycophenolate mofetil (MMF) + Standard dose of cyclosporine (Active Comparator): Patients were treated with 1 gram twice a day (2 grams/day) of Mycophenolate mofetil (MMF) and standard dose of cyclosporine for 12 months post renal transplant. Patients were treated with antibody induction therapy using 20 mg basiliximab two hours prior to transplant and 20 mg basiliximab 4 days post transplant or according to local practice. Corticosteroids were administered according to local practice. Patients were treated for 12 months in the core study and 12 months in the extension study.
  Interventions: Drug: Mycophenolate mofetil (MMF); Drug: Basiliximab; Drug: Cyclosporine A; Drug: Corticosteroid

INTERVENTIONS:
Drug: Everolimus — 0.75 mg twice daily, trough level adjusting between 3 and 8 ng/ml.
  Other Names: Certican
  Arms: Everolimus + Reduced dose of cyclosporine
Drug: Mycophenolate mofetil (MMF) — The initial dose of 2 gm/day Mycophenolate mofetil was started within 24-36 hours from reperfusion after transplantation. MMF was administered daily for 12 months in the core study and 12 months in the extension study.
  Other Names: MMF
  Arms: Mycophenolate mofetil (MMF) + Standard dose of cyclosporine
Drug: Basiliximab — Patients received first dose of basiliximab (20 mg) 2 hours prior to transplantation and 20 mg at Day 4 or according to local practice
Drug: Cyclosporine A — The cyclosporine was initiated either pre-transplant or within 24 hours after transplantation following local regime. Standard dose of cyclosporine was administered with MMF. The Reduced dose of cyclosporine was administered with everolimus.
  Other Names: Neoral®
Drug: Corticosteroid — Corticosteroid was administered according to local practice during the trial but at a dose not less than 5mg per day for 12 months of the study

SUMMARY:
The 12 Month Core Study (CRAD001A1202) was designed to evaluate the efficacy and safety comparing concentration-controlled everolimus (1.5 mg/day starting dose) with reduced dose cyclosporine and corticosteroids versus 2 g/day mycophenolate mofetil (MMF) with standard dose cyclosporine and corticosteroids in de novo renal transplant recipients.

Extension Study (CRAD001A1202E1): Until 24 months after renal transplantation, the study was designed to evaluate the long-term safety and efficacy comparing concentration-controlled everolimus with reduced dose cyclosporine (Neoral®) and corticosteroids versus mycophenolate mofetil with standard dose Neoral® and corticosteroids in de novo renal transplant recipients. Beyond 24 months after renal transplantation, the study was designed to provide everolimus treatment for patients in everolimus group until everolimus is approved and marketed in Japan.

ELIGIBILITY:
Core Study Inclusion Criteria:

* Male or female de novo renal transplant recipients between 18 and 65 years of age
* Patients who are receiving a primary cadaveric donor or non-human leukocyte antigen (non-HLA) identical living donor kidney transplant
* Patients who have given written informed consent to participate in the study
* Females capable of becoming pregnant must have a negative pregnancy test prior to randomization.

Core Study Exclusion Criteria:

* Patients with no evidence of graft function within 24 hours of transplantation are excluded
* Recipients of dual kidney transplants
* Patients who are recipients of multiple solid organ or tissue transplants, or have previously received an organ or tissue transplant.
* Recipients of kidneys from HLA-identical living related donors
* Patients who are recipients of ABO incompatible transplants or T cell cross match positive transplant. Although Panel Reactive Antibodies (PRA) test is not mandatory, patients whose most recent anti-HLA Class I PRA >20% By a CDC-(Complement dependent cytotoxicity) based assay or >50% by a Flow Cytometry or ELISA (Enzyme linked immunosorbent assay) -based assay
* Patients who have tested positive for human immunodeficiency virus (HIV), hepatitis C virus (HCV), or Hepatitis B surface antigen. Laboratory results obtained within 6 months prior to randomization are acceptable, otherwise these tests should be performed within two weeks prior to randomization.
* Recipients of organs from donors who test positive for Hepatitis B surface antigen, HCV or HIV are excluded
* Donor organ with a cold ischemia time >24 hours
* Donor age greater than 65 years
* Patients with platelet count <100,000/mm at baseline before transplantation
* Patients with an absolute neutrophil count of < 1,500/mm³ or white blood cell count of < 4,500/mm³ at baseline before transplantation
* Patients who have severe hypercholesterolemia (>350 mg/dL; >9 mmol/L) or hypertriglyceridemia (>500 mg/dL; >8.5 mmol/L). Patients with controlled hyperlipidemia are acceptable
* Patients who have an abnormal liver profile such as alanine aminotransferase (ALT), Aspartate aminotransferase (AST), alkaline phosphatase (ALP) or total bilirubin >3 times the upper limit of normal (ULN)
* Patients with a known hypersensitivity to either of the study drugs or their class, or to any of the excipients
* Patients who are treated with drugs that are strong inducers or inhibitors of cytochrome P450
* Patients who are unable to take oral medication at time of randomization
* Patients who received an investigational drug or who have been treated with a non-protocol immunosuppressive drug or treatment within 30 days or 5 half-lives prior to randomization
* Patients with a history of malignancy of any organ system, treated or untreated, within the past 5 years whether or not there is evidence of local recurrence or metastases, with the exception of localized excised non-melanomatous skin lesions
* Patients with clinically significant systemic infection at time of transplant or within two weeks prior to transplant
* Patients with a history of severe diarrhea, active peptic ulcer disease, or uncontrolled diabetes mellitus
* Patients who have cardiac failure at time of screening (resting dyspnea, with Grade ≥ 3 according to Old New York Heart Association Classification (Appendix 7) or any severe cardiac disease as determined by the investigator
* Patients who have any surgical or medical condition, which in the opinion of the investigator, might significantly alter the absorption, distribution, metabolism and excretion of study medication
* Patients with abnormal physical or laboratory findings of clinical significance within 2 weeks prior to randomization which would interfere with the objectives of the study
* Patients with any history of coagulopathy or medical condition requiring long-term anticoagulation which would preclude renal biopsy after transplantation. (Low dose aspirin treatment or interruption of chronic anticoagulant is allowed)
* Females of childbearing potential who are planning to become pregnant, who are pregnant and/or lactating, who are unwilling to use effective means of contraception.

Extension Study Inclusion Criteria:

* Patients who completed Month 12 visit in core study (including patients who had discontinued study medication)
* Patients who had given written informed consent to participate in this extension study

Extension Study Exclusion Criteria:

* Women of childbearing potential who were planning to become pregnant, who were unwilling to use two or more effective means of contraception, including abstinence judged by the investigator, surgical sterilization (e.g. bilateral tubal ligation, hysterectomy), hormonal contraception (implantable, patch, oral), and barrier methods (male or female condom with spermicidal gel, diaphragm, sponge, cervical cap). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal were not acceptable methods of contraception.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2008-02; Primary Completion 2010-08 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Novartis Pharma K.K., Japan, Tokyo, Japan

REFERENCES:
- [Derived] Takahashi K, Uchida K, Yoshimura N, Takahara S, Teraoka S, Teshima R, Cornu-Artis C, Kobayashi E. Efficacy and safety of concentration-controlled everolimus with reduced-dose cyclosporine in Japanese de novo renal transplant patients: 12-month results. Transplant Res. 2013 Jul 16;2(1):14. doi: 10.1186/2047-1440-2-14. PMID 23866828

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Core Study randomization was conducted within 24 hours post reperfusion. Participants who completed the 12 month visit of the Core Study and met inclusion/exclusion criteria were eligible to participate in the Extension Study and continued the same treatment as the Core Study until Month 24.
Period: Core Study: 12 Months
Arm/Group | Everolimus + Reduced Dose of Cyclosporine | Mycophenolate Mofetil (MMF) + Standard Dose of Cyclosporine
Started | 61 | 61
Completed | 56 | 58
Not Completed | 5 | 3
Not completed — Subject withdrew consent | 5 | 3
Period: Extension Study: Month 12 to Month 24
Arm/Group | Everolimus + Reduced Dose of Cyclosporine | Mycophenolate Mofetil (MMF) + Standard Dose of Cyclosporine
Started | 53 | 57
Extension ITT: Received Study Drug | 50 | 50
Completed | 47 | 50
Not Completed | 6 | 7
Not completed — Subject withdrew consent | 3 | 0
Not completed — Did not receive study drug in Extension | 3 | 7
Period: Extension Study: After Month 24
Arm/Group | Everolimus + Reduced Dose of Cyclosporine | Mycophenolate Mofetil (MMF) + Standard Dose of Cyclosporine
Started | 44 | 0
Completed | 42 | 0
Not Completed | 2 | 0
Not completed — Subject withdrew consent | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Measures are based on the data obtained in the Core Study.
Groups:
- Everolimus + Reduced Dose of Cyclosporine: An initial everolimus dose of 0.75 mg orally twice daily (1.5 mg/day) was administered 24-36 hours from reperfusion after transplantation and dose adjustments based on everolimus trough level (target trough level 3-8ng/mL).Reduced dose of cyclosporine was initiated either pre-transplantation or within 24 hours after transplantation following the local regimen. Patients were treated with antibody induction therapy using 20 mg basiliximab two hours prior to transplant and 20 mg basiliximab 4 days post transplant or according to local practice. Corticosteroids were administered according to local practice.
- Mycophenolate Mofetil (MMF) + Standard Dose of Cyclosporine: Patients were treated with 1 gram twice a day (2 grams/day) of Mycophenolate mofetil (MMF) and standard dose of cyclosporine for 12 months post renal transplant. Patients were treated with antibody induction therapy using 20 mg basiliximab two hours prior to transplant and 20mg basiliximab 4 days post transplant or according to local practice. Corticosteroids were administered according to local practice.
- Total: Total of all reporting groups
Arm/Group | Everolimus + Reduced Dose of Cyclosporine | Mycophenolate Mofetil (MMF) + Standard Dose of Cyclosporine | Total
Number analyzed (Participants) | 61 | 61 | 122
Age Continuous [Mean (Standard Deviation); unit: years] | 42.5 (14.13) | 38.6 (11.36) | 40.5 (12.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 24 | 39
  Male | 46 | 37 | 83

OUTCOME MEASURES:

1. Primary Outcome: Core Study: Number of Patients With Composite Efficacy Endpoint
Description: The composite efficacy endpoint consisted of treated biopsy proven acute rejection (BPAR) episodes, graft loss, death or loss to follow-up. A treated BPAR was defined as a biopsy graded IA, IB, IIA, IIB, or III and which was treated with anti-rejection therapy. The allograft was presumed to be lost on the day the patient starts dialysis and was not able to stop dialysis. If the patient underwent a graft nephrectomy, then the day of nephrectomy was considered as the day of graft loss.
  For the individual components (including loss of follow-up)of the composite endpoint, patients are counted for the first event to occur.
Time Frame: 12 months
Population: The Intent-To-Treat (ITT) population consisted of all patients randomized after transplantation.
Measure: Number; unit: Participants
Arm/Group | Everolimus + Reduced Dose of Cyclosporine | Mycophenolate Mofetil (MMF) + Standard Dose of Cyclosporine
Number analyzed (Participants) | 61 | 61
Participants
  Composite Efficacy Endpoint | 7 | 7
  Treated BPAR | 3 | 5
  Graft Loss | 0 | 0
  Death | 0 | 0
  Loss to follow up (see caveats) | 4 | 2

2. Secondary Outcome: Core Study: Number Participants With Combined Graft Loss, Death or Loss to Follow-up
Description: The allograft was presumed to be lost on the day the patient starts dialysis and was not able to stop dialysis. If the patient underwent a graft nephrectomy, then the day of nephrectomy was considered as the day of graft loss.
  A loss to follow-up in graft loss, death or loss to follow-up is a patient who did not experience graft loss or death and whose last day of contact was prior to Day 316, i.e. prior to the Month 12 visit window.
Time Frame: 12 months
Population: The Intent-To-Treat (ITT) population consisted of all patients randomized after transplantation.
Measure: Number; unit: Participants
Arm/Group | Everolimus + Reduced Dose of Cyclosporine | Mycophenolate Mofetil (MMF) + Standard Dose of Cyclosporine
Number analyzed (Participants) | 61 | 61
Participants | 5 | 3

3. Secondary Outcome: Core Study: Renal Function Measured by Calculated Glomerular Filtration Rate (cGFR) Using Modification of Diet in Renal Disease (MDRD) Formula
Description: Modification of Diet in Renal Disease (MDRD) formula is:
  Calculated GFR [mL/min/1.73m^2] = 186.3*(C^-1.154)*(A^-0.203)*G*R where
  * C is the serum concentration of creatinine [mg/dL],
  * A is patient age at sample collection date [years],
  * G=0.742 when gender is female, otherwise G=1,
  * R=1.21 when race is black, otherwise R=1
Time Frame: Month 12
Measure: Median (Full Range); unit: mL/min/1.73m^2
Arm/Group | Everolimus + Reduced Dose of Cyclosporine | Mycophenolate Mofetil (MMF) + Standard Dose of Cyclosporine
Number analyzed (Participants) | 61 | 61
mL/min/1.73m^2 | 58.00 (18.993) [17.8 to 123.3] | 55.25 (15.227) [26.1 to 111.8]

4. Primary Outcome: Extension Study: Renal Function Measured by Calculated Glomerular Filtration Rate (cGFR) Using the Modification of Diet in Renal Disease (MDRD) Formula
Description: Renal function was assessed by glomerular filtration rate (GFR) using the MDRD formula:
  GFR [mL/min/1.73m2] = 186.3*(C-1.154)*(A-0.203)*G*R C is the serum concentration of creatinine [mg/dL] A is age [years] G = 0.742 when gender is female, otherwise G=1 R = 1.21 when race is black, otherwise R=1
  Loss to follow up (in In Primary Core Outcome Measure) is composite efficacy failure and contains incidence of treated BPAR, graft loss, death or loss to follow-up
Time Frame: Month 24
Population: Participants from the Extension Intent-to-treat population with data available for analyses.
Measure: Median (Full Range); unit: mL/min/1.73m^2
Groups:
- Everolimus + Reduced Dose of Cyclosporine: An initial everolimus dose of 0.7 5mg orally twice daily (1.5 mg/day) was administered 24-36 hours from reperfusion after transplantation and dose adjustments based on everolimus trough level (target trough level 3-8 ng/mL). Reduced dose of cyclosporine was initiated either pre-transplantation or within 24 hours after transplantation following the local regimen. Patients were treated with antibody induction therapy using 20 mg basiliximab two hours prior to transplant and 20 mg basiliximab 4 days post transplant or according to local practice. Corticosteroids were administered according to local practice. Patients were treated for 12 months in the core study and 12 months in the extension study. Everolimus was available after 24 months for compassionate use.
- Mycophenolate Mofetil (MMF) + Standard Dose of Cyclosporine: Patients were treated with 1 gram twice a day (2 grams/day) of Mycophenolate mofetil (MMF) and standard dose of cyclosporine for 12 months post renal transplant. Patients were treated with antibody induction therapy using 20 mg basiliximab two hours prior to transplant and 2 0mg basiliximab 4 days post transplant or according to local practice. Corticosteroids were administered according to local practice. Patients were treated for 12 months in the core study and 12 months in the extension study.
Arm/Group | Everolimus + Reduced Dose of Cyclosporine | Mycophenolate Mofetil (MMF) + Standard Dose of Cyclosporine
Number analyzed (Participants) | 49 | 50
mL/min/1.73m^2 | 58.90 [14.4 to 118.9] | 54.95 [28.3 to 92.7]

5. Secondary Outcome: Extension Study: Number of Participants With Combined Efficacy Endpoint: Graft Loss, Death, Loss to Follow-up and/or Treated Biopsy Proven Acute Rejection (BPAR)
Description: Graft loss was defined as the day the patient started dialysis and was not able to subsequently be removed from dialysis or re-transplant.
  Loss-to-follow was a patient who did not experience a treated BPAR, graft loss or death and whose last day of contact was prior to Month 24.
  A Graft Biopsy was done within 48 hours of suspect rejection. Biopsies were read by the local pathologist according to the updated Banff '97 criteria.
  Treated BPAR was based on local laboratory biopsy results and was defined as a biopsy Banff criteria graded IA to III that was treated with anti-rejection therapy.
Time Frame: 24 Months
Population: Extension Intent-to-treat population.
Measure: Number; unit: Participants
Arm/Group | Everolimus + Reduced Dose of Cyclosporine | Mycophenolate Mofetil (MMF) + Standard Dose of Cyclosporine
Number analyzed (Participants) | 50 | 50
Participants
  Combined Efficacy Endpoint | 4 | 5
  Treated BPAR | 3 | 5
  Graft Loss | 0 | 0
  Death | 0 | 0
  Loss to follow-up | 1 | 0

6. Secondary Outcome: Extension Study: Renal Function Measured by Calculated Glomerular Filtration Rate (GFR) Using the Nankivell Formula
Description: The Nankivell formula was used to calculate GFR at Month 24:
  GFR[mL/min]=6.7/C + W/4 - UREA/2 - 100/H^2 + 35 (25 for females) W= body weight [kg] H= height [m] C= serum creatinine [mmol/L] UREA= serum urea [mmol\L]
Time Frame: Month 24, Month 48
Population: Participants from the Extension Intent-to-treat population with data available for analyses.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Everolimus + Reduced Dose of Cyclosporine | Mycophenolate Mofetil (MMF) + Standard Dose of Cyclosporine
Number analyzed (Participants) | 46 | 50
mL/min
  Month 24 | 63.49 (20.479) | 59.24 (13.840)
  Month 48 (9,0) | 60.16 (9.892) | NA (NA) — 0 participants in the Mycophenolate mofetil (MMF) + Standard dose of cyclosporine arm after Week 24.

7. Secondary Outcome: Extension Study: Number of Participants With Adverse Events and Serious Adverse Events
Description: Additional information about Adverse Events can be found in the Adverse Event Section.
Time Frame: 24 Months
Population: Participants from the Extension Safety Population.
Measure: Number; unit: Participants
Arm/Group | Everolimus + Reduced Dose of Cyclosporine | Mycophenolate Mofetil (MMF) + Standard Dose of Cyclosporine
Number analyzed (Participants) | 50 | 50
Participants
  Adverse Events | 50 | 50
  Serious Adverse Events | 30 | 30

8. Secondary Outcome: Extension Study: Everolimus Trough Levels
Description: Blood was collected at all visits after Day 3 for trough (collected 5 minutes before study drug dose) everolimus levels and was analyzed at a central laboratory using liquid chromatography mass spectrometry.
Time Frame: Month 24, Month 48
Population: Participants from the Extension safety population with data available for analyses.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Everolimus + Reduced Dose of Cyclosporine
Number analyzed (Participants) | 45
ng/mL
  Month 24 | 5.258 (1.1170)
  Month 48 (n=8) | 4.408 (0.5986)

9. Secondary Outcome: Extension Study: Cyclosporine Trough Levels
Description: Blood was collected at all visits after Day 3 for trough (collected 5 minutes before study drug dose) cyclosporine levels and was analyzed at a central laboratory using immunoassay.
Time Frame: Month 24, Month 48
Population: Participants from the Extension safety population with data available for analyses.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Everolimus + Reduced Dose of Cyclosporine | Mycophenolate Mofetil (MMF) + Standard Dose of Cyclosporine
Number analyzed (Participants) | 44 | 48
ng/mL
  Month 24 | 54.1 (39.07) | 105.5 (44.16)
  Month 48 (n=7,0) | 34.2 (37.94) | NA (NA) — 0 participants in the Mycophenolate mofetil (MMF) + Standard dose of cyclosporine arm at Week 48.

10. Primary Outcome: Extension Study: Renal Function Measured by Calculated Glomerular Filtration Rate (cGFR) Using the Modification of Diet in Renal Disease (MDRD) Formula
Description: Renal function was assessed by glomerular filtration rate (GFR) using the MDRD formula:
  GFR [mL/min/1.73m2] = 186.3*(C-1.154)*(A-0.203)*G*R C is the serum concentration of creatinine [mg/dL] A is age [years] G = 0.742 when gender is female, otherwise G=1 R = 1.21 when race is black, otherwise R=1
Time Frame: Month 48
Population: Participants from the Extension Intent-to-treat population with data available for analyses.
Measure: Median (Full Range); unit: mL/min/1.73m^2
Arm/Group | Everolimus + Reduced Dose of Cyclosporine | Mycophenolate Mofetil (MMF) + Standard Dose of Cyclosporine
Number analyzed (Participants) | 9 | 0
mL/min/1.73m^2 | 59.80 [36.8 to 72.0] |

ADVERSE EVENTS:
Description: Combined data of adverse events that occurred in the Core and Extension studies.
Arm/Group | Everolimus + Reduced Dose of Cyclosporine | Mycophenolate Mofetil (MMF) + Standard Dose of Cyclosporine
Serious Adverse Events (participants affected / at risk) | 37/61 | 37/61
Other Adverse Events (participants affected / at risk) | 61/61 | 61/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus + Reduced Dose of Cyclosporine (N=61) | Mycophenolate Mofetil (MMF) + Standard Dose of Cyclosporine (N=61)
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Cataract (Eye disorders) | 2 | 0
Cataract nuclear (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 2 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Impaired healing (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 2
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hepatobiliary disease (Hepatobiliary disorders) | 1 | 0
Adenoviral haemorrhagic cystitis (Infections and infestations) | 1 | 0
Adenovirus infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Cystitis viral (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 1 | 11
Cytomegalovirus viraemia (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 4
Herpes zoster (Infections and infestations) | 1 | 2
Mycobacterium avium complex infection (Infections and infestations) | 1 | 0
Pertussis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 2 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia cytomegaloviral (Infections and infestations) | 1 | 0
Renal cyst infection (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 2
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Kidney rupture (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Ureteric anastomosis complication (Injury, poisoning and procedural complications) | 0 | 1
Bacterial test positive (Investigations) | 1 | 0
Blood beta-D-glucan increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 5 | 6
Blood urea increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0
Cytomegalovirus test positive (Investigations) | 2 | 10
HLA marker study positive (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 | 0
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 1 | 0
Glomerulonephritis membranous (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
IgA nephropathy (Renal and urinary disorders) | 1 | 2
Nephropathy toxic (Renal and urinary disorders) | 1 | 1
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 5 | 2
Renal impairment (Renal and urinary disorders) | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 2 | 0
Azoospermia (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 | 0
Angiopathy (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus + Reduced Dose of Cyclosporine (N=61) | Mycophenolate Mofetil (MMF) + Standard Dose of Cyclosporine (N=61)
Anaemia (Blood and lymphatic system disorders) | 2 | 11
Iron deficiency anaemia (Blood and lymphatic system disorders) | 14 | 16
Leukopenia (Blood and lymphatic system disorders) | 5 | 6
Nephrogenic anaemia (Blood and lymphatic system disorders) | 6 | 8
Palpitations (Cardiac disorders) | 4 | 1
Cushingoid (Endocrine disorders) | 2 | 5
Conjunctivitis (Eye disorders) | 4 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 4
Constipation (Gastrointestinal disorders) | 19 | 27
Dental caries (Gastrointestinal disorders) | 5 | 2
Diarrhoea (Gastrointestinal disorders) | 22 | 15
Gastritis (Gastrointestinal disorders) | 5 | 2
Haemorrhoids (Gastrointestinal disorders) | 4 | 2
Nausea (Gastrointestinal disorders) | 9 | 13
Periodontitis (Gastrointestinal disorders) | 5 | 3
Stomatitis (Gastrointestinal disorders) | 15 | 10
Vomiting (Gastrointestinal disorders) | 7 | 7
Generalised oedema (General disorders) | 8 | 5
Impaired healing (General disorders) | 5 | 1
Oedema peripheral (General disorders) | 14 | 5
Pyrexia (General disorders) | 14 | 17
Hepatic function abnormal (Hepatobiliary disorders) | 11 | 4
Cystitis (Infections and infestations) | 3 | 5
Cytomegalovirus infection (Infections and infestations) | 2 | 10
Cytomegalovirus viraemia (Infections and infestations) | 0 | 4
Gastroenteritis (Infections and infestations) | 7 | 2
Nasopharyngitis (Infections and infestations) | 37 | 38
Oral herpes (Infections and infestations) | 6 | 5
Pharyngitis (Infections and infestations) | 4 | 3
Urinary tract infection (Infections and infestations) | 10 | 9
Procedural pain (Injury, poisoning and procedural complications) | 8 | 3
Wound complication (Injury, poisoning and procedural complications) | 9 | 4
Alanine aminotransferase increased (Investigations) | 5 | 6
Blood alkaline phosphatase increased (Investigations) | 13 | 7
Blood creatine phosphokinase increased (Investigations) | 4 | 1
Blood creatinine increased (Investigations) | 10 | 10
Blood follicle stimulating hormone increased (Investigations) | 10 | 1
Blood luteinising hormone increased (Investigations) | 10 | 0
C-reactive protein increased (Investigations) | 4 | 0
Cytomegalovirus test positive (Investigations) | 3 | 16
Low density lipoprotein increased (Investigations) | 4 | 0
Weight increased (Investigations) | 6 | 5
Decreased appetite (Metabolism and nutrition disorders) | 3 | 4
Dehydration (Metabolism and nutrition disorders) | 3 | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 11 | 4
Hypercholesterolaemia (Metabolism and nutrition disorders) | 7 | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 4
Hyperlipidaemia (Metabolism and nutrition disorders) | 30 | 20
Hyperuricaemia (Metabolism and nutrition disorders) | 12 | 15
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 7
Hypophosphataemia (Metabolism and nutrition disorders) | 4 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 16
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 3
Osteoporosis (Musculoskeletal and connective tissue disorders) | 4 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 4
Dizziness (Nervous system disorders) | 0 | 5
Dizziness postural (Nervous system disorders) | 0 | 4
Headache (Nervous system disorders) | 16 | 9
Hypoaesthesia (Nervous system disorders) | 6 | 3
Tremor (Nervous system disorders) | 5 | 1
Insomnia (Psychiatric disorders) | 17 | 9
Bladder irritation (Renal and urinary disorders) | 5 | 3
Dysuria (Renal and urinary disorders) | 4 | 5
Haematuria (Renal and urinary disorders) | 5 | 6
Nephropathy toxic (Renal and urinary disorders) | 13 | 5
Proteinuria (Renal and urinary disorders) | 10 | 5
Tubulointerstitial nephritis (Renal and urinary disorders) | 5 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Acne (Skin and subcutaneous tissue disorders) | 18 | 22
Hirsutism (Skin and subcutaneous tissue disorders) | 1 | 4
Rash (Skin and subcutaneous tissue disorders) | 5 | 1
Hypertension (Vascular disorders) | 21 | 18
Lymphocele (Vascular disorders) | 6 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.